CLINICAL TRIAL: NCT01951885
Title: Tacrolimus, Mini-dose Methotrexate and Mycophenolate Mofetil Versus Tacrolimus and Methotrexate for the Prevention of Acute Graft-versus-Host-Disease
Brief Title: Tac, Mini-MTX, MMF Versus Tac, MTX for GVHD Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6Z13
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Acute Biphenotypic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Hodgkins Disease; Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — Tacrolimus; Methotrexate; merphos; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (tacrolimus, methotrexate) (Active Comparator): Participants receive tacrolimus IV over 24 hours beginning on day -1 (or tacrolimus orally beginning on day -3) and then PO BID after engraftment with a taper from day 100 to day 180 (in the absence of GVHD). Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Drug: tacrolimus; Drug: methotrexate
- Group B (tacrolimus, methotrexate, mycophenolate mofetil) (Experimental): Patients receive tacrolimus as in group A and methotrexate (low dose) IV on days 1, 3, and 6. Patients also receive oral mycophenolate mofetil BID beginning on day 1, with a taper from day 45 to day 100 (in the absence of GVHD).
  Interventions: Drug: tacrolimus; Drug: Mycophenolate mofetil; Drug: Methotrexate (low dose)

INTERVENTIONS:
Drug: tacrolimus — Tacrolimus 0.03 mg/kg/day beginning day -1 or tacrolimus 0.03mg/kg/dose BID orally beginning on day -3. If Tac is administered intravenously, it will be given over 24 hours and will be converted to oral administration 2 times a day when the patient has engrafted and/or can tolerate oral medication. Levels of Tac will be obtained to maintain a recommended target serum level of 5-12 ng/mL
  Other Names: FK 506; Prograf
Drug: methotrexate — MTX 15mg/m2 IV on day +1, followed by 10mg/m2 on day +3, +6, +11. If patient < 10 kg then MTX will be given at 0.5 mg/kg IV on day +1. Then MTX will be given at 0.33 mg/kg on days +3, +6 and +11.
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Group A (tacrolimus, methotrexate)
Drug: Mycophenolate mofetil — Patients will receive Mycophenolate beginning on day +1. Patients >40 kg will receive Mycophenolate 1000 mg twice a day. Mycophenolate should be given orally twice a day. IV formulation may be used if the patient cannot tolerate oral route. Patients < 40 kg will receive MMF 45 mg/kg/day (15 mg/kg three times a day). MMF may be given orally or intravenously as per institutional protocol
  Other Names: Cellcept; MMF
  Arms: Group B (tacrolimus, methotrexate, mycophenolate mofetil)
Drug: Methotrexate (low dose) — MTX 5mg/m2 IV on day +1, +3, +6. If patient<10 kg MTX will be given at 0.17 mg/kg on day +1, +3, and +6.
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Group B (tacrolimus, methotrexate, mycophenolate mofetil)

SUMMARY:
This randomized clinical trial studies standard GVHD prophylaxis with tacrolimus and methotrexate compared to tacrolimus, mycophenolate mofetil and a reduced-dose methotrexate in patients with hematologic malignancies undergoing allogeneic hematopoietic cell transplant. Both mycophenolate mofetil and reduced-dose methotrexate, in combination with a calcineurin inhibitor, have been shown to be safe and effective in GVHD prevention with less toxicity than standard dose methotrexate. It is not yet known, however, whether this combination of mycophenolate mofetil and reduced-dose methotrexate with tacrolimus is more effective than tacrolimus and standard dose methotrexate in preventing GVHD.

DETAILED DESCRIPTION:
Study Design This is a prospective randomized trial to determine the effectiveness of different doses of GVHD prophylaxis on mucositis, engraftment and aGVHD. Study consists of two study groups of 50 subjects each.

Group A will receive Tac and MTX (15 mg/m2 day +1, 10 mg/m2 day +3, +6, +11). Group B will receive Tac, Mini-dose MTX (5 mg/m2 on day +1, +3, +6) and MMF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following documented diseases:

  * Chronic myelogenous leukemia
  * Chronic lymphocytic leukemia
  * Multiple myeloma
  * Myelodysplasia
  * Myeloproliferative disorder
  * Non-Hodgkin's lymphoma
  * Hodgkin's disease
  * Acute myelogenous leukemia
  * Acute lymphoblastic leukemia
  * Acute biphenotypic leukemia
* Patients must be undergoing a myeloablative allogeneic hematopoietic cell transplant with one of the following conditioning regimens:

  * Busulfan (≥ 12.8 mg/kg IV or PO) and cyclophosphamide (≥ 120 mg/kg)

    --- Busulfan dose may be adjusted according to pharmacokinetics targeting a daily AUC of 5000 μmol-min/L, per institution standard of practice.
  * Total body irradiation (TBI) (≥ 1200 cGy) and etoposide (60 mg/kg)
  * TBI (≥ 1200 cGy) and cyclophosphamide (120 mg/kg)
* Patient must have achieved and be in complete morphologic remission prior to starting conditioning regimen
* Patient's donor must be a related or unrelated human leukocyte antigen (HLA) 8/8 allele-level match (HLA-A, B, C and DRB1)
* Adult patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; pediatric patients must have Lansky score ≥ 60%
* Patients must have a life expectancy of 100 days
* Patients must sign written informed consent

Exclusion Criteria:

* Patients who have undergone any prior transplant
* Patients who are seropositive for human immunodeficiency virus (HIV)
* Patients with any medical illness or concurrent psychiatric illness which, in the investigators' opinion, cannot be adequately controlled with appropriate therapy
* Patients who are pregnant or lactating

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Hamilton, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Hamilton BK, Rybicki LA, Li H, Lucas T, Corrigan D, Kalaycio M, Sobecks R, Hanna R, Rotz SJ, Dean RM, Gerds AT, Jagadeesh D, Brunstein C, Sauter CS, Copelan EA, Majhail NS. Tacrolimus/methotrexate vs tacrolimus/reduced-dose methotrexate/mycophenolate for graft-versus-host disease prevention. Blood Adv. 2023 Aug 22;7(16):4505-4513. doi: 10.1182/bloodadvances.2023010310. PMID 37352262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from local hospital from July 2014 thru July 2020
Period: Overall Study
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Started | 50 | 51
Completed | 49 | 47
Not Completed | 1 | 4
Not completed — ineligible due to a change in conditioning regimen | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — ineligible due to a change in donor | 0 | 1
Not completed — ineligible after experiencing cardiac issues | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants that went on study
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil) | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Customized [Count of Participants; unit: Participants]
  0-9 years old | 1 | 1 | 2
  10-19 years old | 0 | 3 | 3
  20-29 years old | 10 | 7 | 17
  30-39 years old | 9 | 8 | 17
  40-49 years old | 11 | 12 | 23
  50-59 years old | 19 | 15 | 34
  60-69 years old | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 18 | 46
  Male | 22 | 33 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 47 | 51 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Severe (Grade 3-4) Mucositis Graded According to the World Health Organization (WHO) Grading Scale
Description: Participants (percentage of) will be graded three times per week through day 28 of the study. Incidence will be compared through Wilcoxon rank sum tests.
  The WHO grading scale for mucositis is scaled depending on the severity of mucositis symptoms, with a lower stage associated with a better outcome and greater stages associated with worse outcomes. The staging is as follows:
  Stage 0: None Stage 1 (mild): Oral soreness, erythema Stage 2 (moderate): Oral erythema, ulcers, solid diet tolerated Stage 3 (severe): Oral ulcers, liquid diet only Stage 4 (life-threatening): Oral alimentation impossible
Time Frame: Up to day 28
Population: participants that completed study
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 81.6 | 57.4
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney); 47 patients per arm were needed to detect a 25% improvement in mucositis based on a one-sided test with 5% significance and 80% power

2. Primary Outcome: Time to Neutrophil Engraftment
Description: The number of days to reach a neutrophil count of greater than or equal to 500/ul for three consecutive laboratory values obtained on different days. The day of engraftment will be the first day of the three consecutive laboratory values.
Time Frame: Up to 28 days
Population: participants that were able to engraft neutrophils
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 47 | 47
days | 17 [11 to 27] | 15 [11 to 23]

3. Primary Outcome: Time to Platelet Engraftment
Description: The number of days to reach a platelet count of greater than or equal to 20,000/ul for three consecutive laboratory values obtained on different days, independent of platelet transfusions the prior 7 days. The day of engraftment will be the first day of the three consecutive laboratory values. For cases of delayed engraftment beyond 28 days, results will be recorded once the participant engrafts.
Time Frame: The date the participant engrafts, up to 28 days
Population: participants that were able to engraft platelets
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 27 | 23
days | 27 [16 to 131] | 23 [10 to 112]

4. Primary Outcome: Cumulative Incidence of Participants With Acute GVHD
Description: Acute GVHD by grade will be estimated using cumulative incidence methods and compared using the Gray test.
  A lower clinical grade and/or stage of GVHD corresponds to a better participant outcome and a higher grade corresponds to a worse participant outcome. Grading is as follows:
  Grade 0: No stage 1-4 of any organ Grade 1: Stage 1-2 skin without liver, upper GI, or lower GI involvement. Grade 2: Stage 3 rash and/or stage 1 liver and/or stage 1 upper GI and/or stage 1 lower GI.
  Grade 3: Stage 2-3 liver and/or stage 2-3 lower GI, with stage 0-3 skin and/or stage 0-1 upper GI.
  Grade 4: Stage 4 skin, liver, or lower GI involvement, with stage 0-1 upper GI.
  A greater stage of GVHD involves worsening end-organ involvement and worse participant outcomes based on the skin, liver, lower GI, and upper GI.
Time Frame: Day 7- Day 100
Population: participants who completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants
  Grade 1-4 | 37 [23 to 50] | 47 [32 to 60]
  Grade 2-4 | 27 [15 to 39] | 28 [16 to 41]
  Grade 3-4 | 4 [1 to 12] | 13 [5 to 24]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — Cumulative incidence methods are compared using the Gray test with a p-value <0.05; p < 0.05, Log Rank

5. Secondary Outcome: Length of Hospitalization
Description: Hospital stay will be compared between patients in groups A and B using the Wilcoxon rank sum test.
Time Frame: Date of transplant to date of discharge, assessed up to 1 year
Population: participants who completed the study
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
days | 31 [22 to 89] | 27 [20 to 55]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — Hospital stay will be compared between groups using the Wilcoxon rank sum test with a p value of 0.05; p = 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage of Participants Using Total Parenteral Nutrition (TPN) Within 100 Days
Description: TPN use will be compared using the Chi-square test.
Time Frame: Up to day 100
Population: participants who completed the study
Measure: Number; unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 41 | 38
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — TPN use will be compared using the Chi-square test; p < 0.05, Chi-squared

7. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method and compared between the 2 groups using the log-rank test.
Time Frame: Up to 1 year
Population: participants who completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 71 [56 to 82] | 72 [57 to 83]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — Overall survival was estimated using the Kaplan-Meier method and compared between patients receiving Tac/MTX versus Tac/mini-MTX/MMF using the log-rank test; p < 0.05, Log Rank

8. Secondary Outcome: Progression-free Survival
Description: Estimated using the Kaplan-Meier method and compared between the 2 groups using the log-rank test.
Time Frame: Up to 1 year
Population: participants who completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 59 [44 to 71] | 68 [53 to 79]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — Progression-free survival was estimated using the Kaplan-Meier method and compared between patients receiving Tac/MTX versus Tac/mini-MTX/MMF using the log-rank test; p < 0.05, Log Rank

9. Secondary Outcome: Incidence of Chronic GVHD
Description: Chronic GVHD will be graded as mild, moderate, or severe based on the National Institutes of Health Consensus Development Project. The type and duration of immunosuppressive treatment given for cGVHD will be recorded. Mild grades are associated with a better participant outcome and severe corresponds to a worse participant outcome. Grading is as follows:
  Mild: 1 or 2 organs involved with no more than score 1 plus Lung score 0
  Moderate: 3 or more organs involved with no more than score 1 OR At least 1 organ (not lung) with a score of 2 OR Lung score 1
  Severe: At least 1 organ with a score of 3 OR Lung score of 2 or 3
  Organ scores can range from 0 to 3, with 0 being no symptoms on the target organ and a better participant outcome while a score of 3 correlates to severe symptoms on the target organ and worse participant outcomes.
  Potential target organs include: skin, mouth, eyes, GI tract, liver, lungs, joint /fascia, and genital tract
Time Frame: at 6 months
Population: participants who completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants
  any chronic GVHD | 16 [8 to 28] | 15 [6 to 27]
  moderate-severe chronic GVHD | 12 [5 to 23] | 11 [4 to 21]

10. Secondary Outcome: Incidence of Chronic GVHD
Description: as for outcome 9
Time Frame: at 12 months
Population: participants who completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants
  any chronic GVHD | 25 [13 to 37] | 36 [23 to 50]
  moderate-severe chronic GVHD | 20 [10 to 33] | 23 [12 to 36]

11. Secondary Outcome: Length of Time on Continuous Infusion Narcotics
Description: Start and stop dates for the need of continuous IV infusion of narcotics for severe mucositis pain will be recorded. Time on IV infusion will be compared between patients in groups A and B using the Wilcoxon rank sum test.
Time Frame: up to +28 day
Population: Participants that were on continuous infusion narcotics
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
days | 10 [1 to 19] | 9 [2 to 25]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — Infusion times will be compared using the Wilcoxon rank sum test; p < 0.05, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Incidence of Infection
Description: 100-day incidence of infection will be compared using a the Gray test.
Time Frame: Up to day +100
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 63 [48 to 75] | 53 [38 to 66]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 100-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

13. Secondary Outcome: Incidence of Hepatotoxicity as Measured by Bilirubin
Description: 100-day incidence of hepatotoxicity will be compared using a Gray test. Median and range of largest total bilirubin (mg/dL),
Time Frame: Up to day +100
Population: participants that completed the study
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
mg/dL | 1.5 [0.4 to 45.2] | 1.1 [0.4 to 43.8]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 100-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

14. Secondary Outcome: Incidence of Hepatotoxicity as Measured by Elevated Liver Enzymes
Description: 100-day incidence of hepatotoxicity will be compared using a Gray test. Percentage of patients with elevated Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and alkaline phosphatase and a 95% confidence interval
Time Frame: Up to day +100
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants
  AST | 29 [17 to 43] | 15 [6 to 28]
  ALT | 33 [20 to 48] | 28 [16 to 43]
  Alkaline Phosphatase | 2 [0 to 11] | 2 [0 to 11]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 100-day incidence of complications will be compared using the Gray test; p < 0.05, Chi-squared

15. Secondary Outcome: Incidence of Hepatotoxicity as Measured by Veno-occlusive Disease (VOD)
Description: 100-day incidence of hepatotoxicity will be compared using the Gray test. Percentage of patients with VOD and 95% confidence interval
Time Frame: Up to day +100
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 8 [2 to 20] | 2 [0 to 11]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 100-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

16. Secondary Outcome: Incidence of Nephrotoxicity
Description: 100-day incidence of nephrotoxicity will be compared using a Chi-squared test. Percentage of patients requiring dialysis and those with elevated creatinine using a 95% confidence interval
Time Frame: Up to day +100
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants
  Participants requiring dialysis | 12 [5 to 25] | 4 [1 to 15]
  Participants with elevated creatinine | 27 [15 to 41] | 2 [0 to 11]

17. Secondary Outcome: Incidence of Pulmonary Toxicity Measured by Pulmonary Hemorrhage
Description: 180-day incidence of pulmonary toxicity will be compared using the Gray test. Percentage of patients with pulmonary hemorrhage and 95% confidence interval
Time Frame: Up to day +180
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 2 [0 to 11] | 2 [0 to 11]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 180-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

18. Secondary Outcome: Incidence of Pulmonary Toxicity Measured by Pulmonary Edema
Description: 180-day incidence of pulmonary toxicity will be compared using the Gray test. Percentage of patients with pulmonary edema and 95% confidence interval
Time Frame: Up to day +180
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 14 [6 to 27] | 4 [1 to 15]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 180-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

19. Secondary Outcome: Incidence of Pulmonary Toxicity Measured by Respiratory Failure
Description: 180-day incidence of pulmonary toxicity will be compared using the Gray test. Percentage of patients with respiratory failure and 95% confidence interval
Time Frame: Up to day +180
Population: participants that completed the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
Number analyzed (Participants) | 49 | 47
percentage of participants | 9 [4 to 15] | 6 [1 to 8]
Statistical Analysis 1: Comparison: Group A (Tacrolimus, Methotrexate) vs Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil); Test type: Non-Inferiority — 180-day incidence of complications will be compared using the Gray test; p < 0.05, Gray Test

20. Other Pre Specified Outcome: Chimerism Results
Description: Donor chimerism will be assessed by analysis of single-tandem repeats on whole marrow and in lymphocyte enriched or sorted CD3+ T cells and CD33+ granulocytes. Blood will be obtained for donor chimerism "Bone Marrow Engraftment analysis" at approximately 1, 2, 3, 6, 9 and 12 months or as clinically indicated.
Time Frame: Up to one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through one year post transplant
Arm/Group | Group A (Tacrolimus, Methotrexate) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil)
All-Cause Mortality (participants affected / at risk) | 25/50 | 15/51
Serious Adverse Events (participants affected / at risk) | 13/50 | 3/51
Other Adverse Events (participants affected / at risk) | 49/50 | 47/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Tacrolimus, Methotrexate) (N=50) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil) (N=51)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (4) | 0 (0)
Escherichia Coli (E-Coli) (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Tacrolimus, Methotrexate) (N=50) | Group B (Tacrolimus, Methotrexate, Mycophenolate Mofetil) (N=51)
abdominal pain (Gastrointestinal disorders) | 26 | 24
diarrhea (Gastrointestinal disorders) | 41 | 43
dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 15
encephalopathy (Nervous system disorders) | 6 | 3
febrile neutropenia (Blood and lymphatic system disorders) | 14 | 11
fever (General disorders) | 33 | 24
hyperglycemia (Metabolism and nutrition disorders) | 9 | 9
hypertension (Vascular disorders) | 22 | 13
hypokalemia (Metabolism and nutrition disorders) | 12 | 14
hypomagnesemia (Metabolism and nutrition disorders) | 26 | 33
hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 1
nausea (Gastrointestinal disorders) | 48 | 44
peripheral motor neuropathy (Nervous system disorders) | 0 | 1
peripheral sensory neuropathy (Nervous system disorders) | 4 | 6
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 5
sepsis (Infections and infestations) | 8 | 3
tremor (Nervous system disorders) | 7 | 8
vomiting (Gastrointestinal disorders) | 43 | 39
Infections and infestations - Other, specify: BK virus (Infections and infestations) | 1 | 8
Infections and infestations - Other, specify: Candida krusei (Infections and infestations) | 2 | 0
Infections and infestations - Other, specify: Clostridioides difficile (Infections and infestations) | 8 | 8
Infections and infestations - Other, specify: Cellulitis (Infections and infestations) | 2 | 0
Infections and infestations - Other, specify: Citrobacter freundii (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Cytomegalovirus (Infections and infestations) | 4 | 6
Infections and infestations - Other, specify: Coronavirus HKU1 (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: COVID-19 (Infections and infestations) | 2 | 0
Infections and infestations - Other, specify: Escherichia coli (Infections and infestations) | 4 | 2
Infections and infestations - Other, specify: Enterobacter cloacae complex (Infections and infestations) | 2 | 1
Infections and infestations - Other, specify: Enterococcus faecalis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Herpes stomatitis (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Herpes zoster (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Influenza A (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Influenza B (Infections and infestations) | 1 | 1
Infections and infestations - Other, specify: Klebsiella oxytoca (Infections and infestations) | 3 | 1
Infections and infestations - Other, specify: Klebsiella pneumoniae (Infections and infestations) | 4 | 0
Infections and infestations - Other, specify: Methicillin-resistant Staphylococcus aureus (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Methicillin-resistant Staphylococcus epidermidis (Infections and infestations) | 6 | 0
Infections and infestations - Other, specify: Pulmonary aspergillosis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Pulmonary mucormycosis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Raoultella species (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Rhinovirus (Infections and infestations) | 1 | 2
Infections and infestations - Other, specify: Respiratory syncytial virus (Infections and infestations) | 0 | 2
Infections and infestations - Other, specify: Sphingomonas (pseudomonas) paucimobilis (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Staphylococcus aureus pneumonia (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Staphylococcus epidermidis (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Streptococcus mitis (Infections and infestations) | 0 | 2
Infections and infestations - Other, specify: Streptococcus mitis oralis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Thrush (Infections and infestations) | 9 | 7
urinary tract infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Varicella zoster (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: Vancomycin-resistant enterococci (Infections and infestations) | 1 | 0
catheter related infection (Infections and infestations) | 0 | 2
abdominal distension (Gastrointestinal disorders) | 1 | 3
acute kidney injury (Renal and urinary disorders) | 24 | 10
adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
agitation (Psychiatric disorders) | 2 | 1
allergic reaction (Immune system disorders) | 0 | 2
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
anal fistula (Gastrointestinal disorders) | 0 | 1
anal pain (Gastrointestinal disorders) | 1 | 0
anal ulcer (Gastrointestinal disorders) | 0 | 2
anemia (Blood and lymphatic system disorders) | 22 | 23
anorexia (Metabolism and nutrition disorders) | 16 | 15
anxiety (Psychiatric disorders) | 16 | 11
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
atrial fibrillation (Cardiac disorders) | 5 | 1
avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 7 | 12
bladder infection (Infections and infestations) | 0 | 1
bloating (Gastrointestinal disorders) | 0 | 3
blurred vision (Eye disorders) | 6 | 3
bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
cardiac arrest (Cardiac disorders) | 1 | 0
chills (General disorders) | 6 | 9
cholecystitis (Hepatobiliary disorders) | 5 | 0
cholesterol high (Investigations) | 0 | 1
colitis (Gastrointestinal disorders) | 2 | 0
confusion (Psychiatric disorders) | 4 | 2
conjunctivitis (Eye disorders) | 2 | 2
constipation (Gastrointestinal disorders) | 25 | 23
cough (Respiratory, thoracic and mediastinal disorders) | 20 | 24
CPK increased (Investigations) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 1 | 3
delirium (Psychiatric disorders) | 10 | 1
depressed level of consciousness (Nervous system disorders) | 1 | 0
depression (Psychiatric disorders) | 7 | 5
dizziness (Nervous system disorders) | 7 | 14
dry eye (Eye disorders) | 6 | 4
dry mouth (Gastrointestinal disorders) | 10 | 10
dry skin (Skin and subcutaneous tissue disorders) | 6 | 6
dysesthesia (Nervous system disorders) | 1 | 1
dysgeusia (Nervous system disorders) | 6 | 4
dyspareunia (Reproductive system and breast disorders) | 2 | 0
dyspepsia (Gastrointestinal disorders) | 3 | 4
dysphagia (Gastrointestinal disorders) | 5 | 7
ear pain (Ear and labyrinth disorders) | 2 | 1
edema cerebral (Nervous system disorders) | 0 | 1
edema face (General disorders) | 9 | 4
edema limbs (General disorders) | 21 | 20
electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 0
enterocolitis (Gastrointestinal disorders) | 1 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 7
erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
FALL (Injury, poisoning and procedural complications) | 4 | 3
FATIGUE (General disorders) | 40 | 35
FECAL INCONTINENCE (Gastrointestinal disorders) | 5 | 4
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 2
FLATULENCE (Gastrointestinal disorders) | 4 | 3
FLOATERS (Eye disorders) | 0 | 1
FLUSHING (Vascular disorders) | 1 | 0
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 2 | 0
FRACTURE (Injury, poisoning and procedural complications) | 1 | 4
GAIT DISTURBANCE (General disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 3 | 1
GASTROPARESIS (Gastrointestinal disorders) | 0 | 1
GENITAL EDEMA (Reproductive system and breast disorders) | 2 | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 9 | 7
GYNECOMASTIA (Reproductive system and breast disorders) | 0 | 1
HALLUCINATIONS (Psychiatric disorders) | 5 | 2
HEADACHE (Nervous system disorders) | 28 | 30
HEMATOMA (Vascular disorders) | 1 | 4
HEMATURIA (Renal and urinary disorders) | 5 | 8
HEMOLYSIS (Blood and lymphatic system disorders) | 3 | 0
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HEMORRHOIDS (Gastrointestinal disorders) | 12 | 9
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HOT FLASHES (Vascular disorders) | 3 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERKALEMIA (Metabolism and nutrition disorders) | 5 | 8
HYPERNATREMIA (Metabolism and nutrition disorders) | 3 | 1
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATREMIA (Metabolism and nutrition disorders) | 10 | 3
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 | 2
HYPOTENSION (Vascular disorders) | 18 | 13
HYPOTHERMIA (General disorders) | 1 | 1
INFUSION RELATED REACTION (General disorders) | 1 | 2
INR INCREASED (Investigations) | 4 | 3
INSOMNIA (Psychiatric disorders) | 11 | 20
IRRITABILITY (General disorders) | 1 | 1
joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify: LABIAL PAIN (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other, specify: LABIAL ULCER (Reproductive system and breast disorders) | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 3 | 0
LARYNGEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LARYNGITIS (Infections and infestations) | 1 | 1
Nervous system disorders - Other, specify: INTRACEREBRAL HEMORRHAGE (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 5 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 1
LIBIDO DECREASED (Psychiatric disorders) | 2 | 1
Endocrine disorders - Other, specify: testosterone deficiency (Endocrine disorders) | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1
Blood and lymphatic system disorders - Other, specify: MACROCYTIC ANEMIA (Blood and lymphatic system disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 1
MALAISE (General disorders) | 2 | 2
MANIA (Psychiatric disorders) | 1 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
ALKALOSIS (Metabolism and nutrition disorders) | 2 | 0
MITRAL VALVE DISEASE (Cardiac disorders) | 1 | 0
Psychiatric disorders - Other, specify: MOOD CHANGES (Psychiatric disorders) | 1 | 0
Musculoskeletal and connective tissue disorders - Other, specify: MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 2 | 2
MUSCLE WEAKNESS LEFT-SIDED (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorders - Other, specify: MYOCLONUS (Musculoskeletal and connective tissue disorders) | 2 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Respiratory, thoracic and mediastinal disorders - Other, specify: NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NECK EDEMA (General disorders) | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 13 | 17
Skin and subcutaneous tissue disorders - Other, specify: NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1
Renal and urinary disorders - Other, specify: NOCTURIA (Renal and urinary disorders) | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 2
Renal and urinary disorders - Other, specify: NONOLIGURIC RENAL FAILURE (Renal and urinary disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: ODYNOPHAGIA (Gastrointestinal disorders) | 9 | 8
ORAL DYSESTHESIA (Gastrointestinal disorders) | 2 | 0
Musculoskeletal and connective tissue disorders - Other, specify: OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 6
PALPITATIONS (Cardiac disorders) | 0 | 2
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: PAPULAR RASH (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify: PAPULE (Skin and subcutaneous tissue disorders) | 1 | 0
PARESTHESIA (Nervous system disorders) | 6 | 8
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 2
PERICARDITIS (Cardiac disorders) | 0 | 1
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrointestinal disorders - Other, specify: PERIRECTAL FISSURE (Gastrointestinal disorders) | 0 | 1
PHLEBITIS (Vascular disorders) | 1 | 0
PHOTOPHOBIA (Eye disorders) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 20 | 24
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 3
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify: PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, specify: PNEUMONIA (Infections and infestations) | 6 | 6
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PROCTITIS (Gastrointestinal disorders) | 1 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 3
PROTEINURIA (Renal and urinary disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 6 | 11
PSYCHOSIS (Psychiatric disorders) | 1 | 1
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 17 | 25
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 2
RECTAL PAIN (Gastrointestinal disorders) | 10 | 7
Eye disorders - Other, specify: RETINAL HEMORRHAGE (Eye disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 6 | 7
General disorders - Other, specify: RIGORS (General disorders) | 4 | 1
SCALP PAIN (Skin and subcutaneous tissue disorders) | 0 | 1
SINUS PAIN (Nervous system disorders) | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 1
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 | 0
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: SMALL BOWEL ISCHEMIA (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Musculoskeletal and connective tissue disorders - Other, specify: STEROID MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
STOMACH PAIN (Gastrointestinal disorders) | 1 | 0
STROKE (Nervous system disorders) | 1 | 0
Eye disorders - Other, specify: SUBCONJUNCTIVAL HEMORRHAGE (Eye disorders) | 2 | 1
SUICIDAL IDEATIONS (Psychiatric disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 0
Blood antidiuretic hormone abnormal (Investigations) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 14 | 11
Respiratory, thoracic and mediastinal disorders - Other, specify: TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 4 | 4
TINNITUS (Eye disorders) | 0 | 2
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 0
TYPHLITIS (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0
UPPER RESPIRATORY INFECTION (Infections and infestations) | 10 | 7
URINARY FREQUENCY (Renal and urinary disorders) | 2 | 4
Renal and urinary disorders - Other, specify: URINARY HESITANCY (Renal and urinary disorders) | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 3
URINARY RETENTION (Renal and urinary disorders) | 4 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 4
URINARY URGENCY (Renal and urinary disorders) | 1 | 5
URTICARIA (Skin and subcutaneous tissue disorders) | 4 | 2
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 8 | 4
VAGINAL DRYNESS (Reproductive system and breast disorders) | 3 | 1
VAGINAL INFECTION (Infections and infestations) | 0 | 1
VAGINAL INFLAMMATION (Reproductive system and breast disorders) | 1 | 2
Reproductive system and breast disorders - Other, specify: VAGINAL ITCHING (Reproductive system and breast disorders) | 3 | 2
VAGINAL PAIN (Reproductive system and breast disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 8 | 3
VERTIGO (Ear and labyrinth disorders) | 0 | 1
Investigations - Other, specify: VITAMIN D DEFICIENCY (Investigations) | 8 | 7
WATERING EYES (Eye disorders) | 3 | 3
WEIGHT GAIN (Investigations) | 3 | 1
WEIGHT LOSS (Investigations) | 2 | 2
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 4 | 6
WHITE BLOOD CELL DECREASED (Investigations) | 16 | 17
irregular menstruation (Reproductive system and breast disorders) | 0 | 1
Eye disorders - Other, specify: decreased visual acuity (Eye disorders) | 1 | 3
Renal and urinary disorders - Other, specify: dysuria (Renal and urinary disorders) | 8 | 11
Infections and infestations - Other, specify: folliculitis (Infections and infestations) | 2 | 2
General disorders, Other, specify: generalized edema (General disorders) | 4 | 4
Renal and urinary disorders - Other, specify: glucosuria (Renal and urinary disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify: hyperlipidemia (Metabolism and nutrition disorders) | 3 | 2
Metabolism and nutrition disorders - Other, specify: hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: ABSCESS (Infections and infestations) | 1 | 2
Renal and urinary disorders - Other, specify: ACUTE TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
Psychiatric disorders - Other, specify: ALTERED MENTAL STATUS (Psychiatric disorders) | 2 | 0
Eye disorders - Other, specify: ANISOCORIA (Eye disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 3 | 0
Cardiac disorders - Other, specify: CARDIAC MURMUR (Cardiac disorders) | 1 | 0
Musculoskeletal and connective tissue disorders - Other, specify: CERVICAL DISC HERNIATION (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatobiliary disorders - Other, specify: CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify: CHOLESTASIS (Hepatobiliary disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: COLONIC ILEUS (Gastrointestinal disorders) | 1 | 0
Eye disorders - Other, specify: CONJUNCTIVAL HEMORRHAGE (Eye disorders) | 1 | 0
Musculoskeletal and connective tissue disorders - Other, specify: COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: CYSTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: DERMATITIS (Skin and subcutaneous tissue disorders) | 4 | 6
Skin and subcutaneous tissue disorders - Other, specify: ATOPIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: DIAPER DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: SEBORRHEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: SPONGIOTIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: DIFFUSE ALVEOLAR HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: DIVERTICULITIS (Gastrointestinal disorders) | 2 | 0
Musculoskeletal and connective tissue disorders - Other, specify: DYSTONIA (Musculoskeletal and connective tissue disorders) | 0 | 1
Ear and labyrinth disorders - Other, specify: EAR BLEEDING (Ear and labyrinth disorders) | 0 | 1
Metabolism and nutrition disorders - Other, specify: EARLY SATIETY (Metabolism and nutrition disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, specify: GASTROENTERITIS (Infections and infestations) | 1 | 0
Gastrointestinal disorders - Other, specify: GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify: HEMATOCHEZIA (Gastrointestinal disorders) | 1 | 6
Vascular disorders - Other, specify: SUBDURAL HEMATOMA (Vascular disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal and urinary disorders - Other, specify: HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 3
Nervous system disorders - Other, specify: HYPERESTHESIA (Nervous system disorders) | 0 | 1
Metabolism and nutrition disorders - Other, specify: INCREASE IN APPETITE (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify: INDIGESTION (Metabolism and nutrition disorders) | 1 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify: RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: SINUS DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Musculoskeletal and connective tissue disorders - Other, specify: HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal and connective tissue disorders - Other, specify: JAW PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal and connective tissue disorders - Other, specify: SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal and connective tissue disorders - Other, specify: RIB PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal and urinary disorders - Other, specify: HEMORRHAGIC CYSTITIS (Renal and urinary disorders) | 0 | 2
Endocrine disorders - Other, specify: HYPERGONADISM (Endocrine disorders) | 0 | 1
Ear and labyrinth disorders - Other, specify: IMPACTED CERUMEN (Ear and labyrinth disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: RHONCHI (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify: INFARCTION OF SPLEEN (Blood and lymphatic system disorders) | 1 | 0
General disorders - Other, specify: generalized body aches (General disorders) | 2 | 2
General disorders - Other, specify: generalized pain (General disorders) | 0 | 2
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 12 | 11
Vascular disorders - Other, specify: SUBARACHNOID HEMORRHAGE (Vascular disorders) | 2 | 0
Eye disorders - Other, specify: SUPERFICIAL PUNCTATE KERATITIS (Eye disorders) | 1 | 0
Nervous system disorders - Other, specify: FOOT DROP (Nervous system disorders) | 1 | 0
Cardiac disorders - Other, specify: DEMAND ISCHEMIA (Cardiac disorders) | 1 | 0
General disorders - Other, specify: CHEST PAIN (General disorders) | 2 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT01951885/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT01951885/ICF_003.pdf